CLINICAL TRIAL: NCT02253238
Title: Sensor-Assisted Prevention of Dehydration in Head and Neck Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0535; 1R01CA177914-01 (NIH); NCI-2015-00946 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Dehydration; Sensor-based home monitoring; Radiation therapy; RT; XRT; Oropharyngeal cancer; Hypopharyngeal cancer; Nasopharyngeal cancer; Salivary gland cancer; Oral cavity cancer; Questionnaires; Surveys; Quality of life; QOL; Phone calls; Self-monitoring devices; CYberinfrastructure for COmparative effectiveness REsearch; CYCORE; Emergency room visits; ER; Emergency room visits with hospitalization; ERHV
MeSH Terms: conditions — Head and Neck Neoplasms; Dehydration; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Nasopharyngeal Neoplasms; Salivary Gland Neoplasms; Mouth Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (Other): Surveys administered in person or by telephone interview and are audio-recorded.
  Interventions: Behavioral: Quality of Life Survey; Behavioral: Health Management Surveys; Behavioral: Symptoms Surveys
- CYCORE Group + Standard of Care (Experimental): Home use of CYCORE devices (blood pressure monitor, weight scale, electronic tablet, palm-sized plug-in computer).
  Surveys administered in person or by telephone interview and are audio-recorded.
  Interventions: Behavioral: Quality of Life Survey; Behavioral: Health Management Surveys; Other: Monitoring Devices; Behavioral: Symptoms Surveys; Behavioral: Device Usability Survey

INTERVENTIONS:
Behavioral: Quality of Life Survey — Quality of life survey completed at baseline, 7 days after radiation therapy (RT) and at 6 - 8 weeks after RT.
  Other Names: Survey
Behavioral: Health Management Surveys — Confidence in health management survey; completed at baseline and 6 - 8 weeks after RT.
  Other Names: Questionnaires
Other: Monitoring Devices — Home use of CYCORE devices (blood pressure monitor, weight scale, electronic tablet, palm-sized plug-in computer)
  Arms: CYCORE Group + Standard of Care
Behavioral: Symptoms Surveys — Behavioral: Symptoms survey 1; completed at weeks 1, 3, 5, and 7 days after RT, and at 6 - 8 weeks after RT.
  Behaviorial: Symptoms survey 2; completed at baseline, weeks 1, 3, 5, and 7 days after RT, and at 6 - 8 weeks after RT.
Behavioral: Device Usability Survey — Device usability survey; completed at weeks 1, 3, 5, and 7 days after RT.
  Other Names: Questionnaire
  Arms: CYCORE Group + Standard of Care

SUMMARY:
The goal of this research study is to learn if home-use of devices to identify dehydration risk, when added to standard care, will help to lower hospitalizations and emergency room visits (and related costs) in patients with head and neck cancer.

CYCORE is a software-based system that enables comprehensive collection, storage and analysis of information related to cancer research and clinical care. In this study, those in the CYCORE group use devices at home to measure their dehydration risk. This information is monitored by their clinicians. Those in the standard care group complete health based surveys, as do those in the CYCORE group.

DETAILED DESCRIPTION:
Abstract:

While head and neck cancer (HNC) is highly curable, primary radiation treatment (RT) is nonetheless challenging. Despite intensive, high-quality, multidisciplinary symptom management of HNC patients during RT, up to 80% of these patients experience moderate to severe levels of oral mucositis making it nearly impossible to drink sufficient fluids and necessitating opioid care for pain. Our data show that 27 - 32% of HNC patients are admitted to inpatient or emergency room (ER) units during RT. Those admissions related to dehydration (and the accompanying costs) are largely preventable, provided at-risk patients can be identified early for intravenous fluid rehydration. Currently, given standard of care for HNC patients undergoing RT, clinicians assess patients only once per week during standard clinic visits. However, the physiological changes underlying the onset of dehydration can develop rapidly, often between clinic visits. In the proposed project, we focus on this missed opportunity for prevention by testing the efficacy of a novel method for home-based dehydration assessment and early intervention to reduce dehydration risk.

This project assesses the efficacy of a coordinated dehydration prevention program using a system (CYCORE) that links home-based monitoring sensors--that collect biometric and self-reported symptom data--to a cyber-infrastructure (CI) and sends these data daily to the patient's healthcare team, who in turn monitor the patients for early signs of dehydration and provide earlier clinical intervention, when needed. The project is based on our successful pilot study that evaluated the feasibility of CYCORE use in HNC patients and with their radiology healthcare team. The patients reported high acceptability of the system, while clinicians perceived the data as valuable and useful in providing additional information regarding patient's at-home dehydration status. We will randomize a total of 192 HNC patients receiving RT at MD Anderson Cancer Center (MDACC) to either standard care or CYCORE + standard care (CYCORE). We hypothesize that patients randomized to CYCORE will experience fewer hospitalizations and ER admissions (and fewer associated costs) due to dehydration compared with patients in the standard care arm.

To the best of our knowledge, the application of a system such as CYCORE has not been explored in the HNC population. Objective, home-based monitoring may be an optimal method of capturing data critical to early evaluation of dehydration risk; other methods, such as patient self-report, are limited by the patient's ability to accurately recall symptoms. MDACC is an ideal environment for conducting the proposed study; more HNC patients are treated with RT at MDACC compared with any other center in Texas, and it is possible to track outcomes and cost-related data, given the HNC patients receive all of their RT-related care, including related hospitalization and ER admissions, at one center. If our efficacy study proves successful, this dehydration prevention model can potentially be applied to other health conditions and in other settings.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of any of the following cancers: stage 1-4b (includes 4a) oropharyngeal, hypopharyngeal, nasopharyngeal, salivary gland or oral cavity; stage 3-4b (includes 4a) laryngeal; any unknown primary head and neck cancer with cervical metastasis that will be addressed with treatment to bilateral necks and mucosa; any thyroid cancer that will be addressed with treatment to the bilateral necks; or other head and neck cancers medically approved by one of our Radiation Oncology collaborating MDs
2. Currently receiving (or scheduled to receive) radiation treatment for a cancer listed in the inclusion criteria
3. Age 18 years or older
4. Fluent in English
5. Radiation treatment for this cancer was completed (or will be completed) at MD Anderson Cancer Center (Post-RT study only)
6. Receiving radiation treatment for this cancer at any site within the MDACC Cancer Network (Cancer Network study only)

Exclusion Criteria:

1. Overt cognitive difficulty demonstrated by not being clearly oriented to person or place or time
2. Zubrod Performance Status >2, or self-reports either not being up and about more than 50% of waking hours or unable to provide self-care
3. History of current oropharyngeal dysphagia unrelated to cancer diagnosis (e.g. dysphagia due to underlying neurogenic disorder)
4. Orthopedic, neurologic, or musculoskeletal disability that would interfere with the functional task of standing on a weight scale
5. Scheduled to receive or receiving unilateral radiation treatment for this cancer
6. Received previous radiation treatment for head and neck cancer
7. Consented to enroll in a trial with a toxicity endpoint
8. Undergoing only palliative (not curative) radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison Between the Two Groups of the Number of Hospitalizations and ER Visits Due to Dehydration | 12 - 15 weeks
  Primary outcome is proportion of patients who experience ER visits and/or hospitalizations related to dehydration (ERV) combined with ER visits resulting in hospitalization through the 6-7 weeks of RT. Primary analysis is comparison of proportion of patients in CYCORE group who have an ERV or ERHV and proportion of patients in the standard care group who have an ERV or ERHV. Analysis consists of a binomial test of two proportions using a continuity-corrected chi-square test. Analyses will follow the intention-to-treat principle, that is a patient in either arm who drops out is assumed to have an ERV and/or ERHV. For comparison purposes, data will be analyzed only using patients who have completed the study.

CONTACTS AND LOCATIONS:
Overall Officials: Susan K. Peterson, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org